CLINICAL TRIAL: NCT02648061
Title: Transitions Between Clinical Circulatory States After Out-of-hospital Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/1807
Record Dates: First submitted 2015-12-04; First posted 2016-01-06 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Out-of-Hospital Cardiac Arrest
Keywords: Blood circulation; Follow-up studies; Biological markers; Hemodynamics
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- After cardiac arrest syndrome (ACAS): adult patients after out-of-hospital cardiac arrest

SUMMARY:
Extensive research exists for cardio-pulmonary resuscitation (CPR) and the chance of successful return of spontaneous circulation (ROSC) is improved. Unfortunately, the overall prognosis after ROSC has not improved much and the in-hospital mortality is still reported to be 50 to 70 %. The "post-resuscitation disease" is now called the "post-cardiac arrest syndrome" (PCAS) and comprises 1) brain injury, 2) myocardial dysfunction and 3) systemic ischemia and reperfusion.

Treatment of patients after cardiac arrest has often followed guidelines that were primarily developed for treatment of septic shock. It is still uncertain whether this is the optimal way to deliver circulatory support after cardiac arrest.

There is a lack of studies assessing the relationship between the inflammatory response measured by inflammatory biomarkers and circulatory failure in PCAS.

In this study a detailed description will be given of the clinical trajectory of the circulation and the inflammatory response during the first 5 days after cardiac arrest, and it will be investigated whether patterns of circulatory and inflammatory response may be predictive of deterioration of clinical state.

DETAILED DESCRIPTION:
This study will obtain longitudinally advanced hemodynamic observations with high resolution during the acute phase of post cardiac arrest syndrome (PCAS), and analyze the details in clinical transitions related to circulatory failure. The study will also analyze the relationship between inflammatory biomarkers and circulatory failure in PCAS and kinetics of hemodynamics associated with standard interventions in the intensive care unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

* Return of spontaneous circulation (ROSC) after out-of-hospital cardiac arrest (OHCA)
* Admitted to Coronary Care Unit (CCU) or Intensive Care Unit (ICU), St. Olav's University Hospital

Exclusion Criteria:

* Sepsis within 24 hours before cardiac arrest
* Pregnancy
* Decision of withdrawal or withholding of life prolonging therapy (i.e. due to advanced malignancy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who are admitted to either the Intensive Care Unit (ICU) or the Coronary Care Unit (CCU) at St. Olav's University Hospital, Trondheim, Norway, after out-of-hospital cardiac arrest will be considered for inclusion.(catchment population of 700,000)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Time in clinical circulatory state (stable, unstable, severe unstable) | 5 days
  These clinical circulatory states are defined as follows: 1) Stable circulation (Mean blood pressure > 65 mmHg, heart rate 51-100, lactate serum concentrations < 2 mmol/l, ScvO2 > 65, fluid administration < 0.5 l/h, norepinephrine dose < 0.1 microgram/kg/min, no other vasoactive drugs.
  2) Unstable circulation (mean blood pressure 45-64 mmHg , heart rate 41-50, 101-130, lactate serum concentrations 2-4 mmol/l, ScvO2 > 50-64, fluid administration 0.5-1,9 l/h, norepinephrine dose 0.1-0.29 microgram/kg/min, Dobutamin > 10 microgram/kg/min, no other vasoactive drugs) 3) Severe unstable circulation (mean blood pressure < 45 mmHg , heart rate < 40, > 130, lactate serum concentrations >4 mmol/l, ScvO2 < 50, fluid administration > 2.0 l/h, norepinephrine dose 0.3 or above microgram/kg/min, dobutamin > 10 microgram/kg/min, other vasoactive drugs, use of aortic balloon pump).

SECONDARY OUTCOMES:
Interleukin-6 in relation to dose of Norepinephrine used to correct vasoplegia after cardiac arrest | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Toril Hernes, prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- St Olavs Hospital Trondheim University Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langeland H, Bergum D, Loberg M, Bjornstad K, Damas JK, Mollnes TE, Skjaervold NK, Klepstad P. Transitions Between Circulatory States After Out-of-Hospital Cardiac Arrest: Protocol for an Observational, Prospective Cohort Study. JMIR Res Protoc. 2018 Jan 19;7(1):e17. doi: 10.2196/resprot.8558. PMID 29351897
- [Result] Langeland H, Bergum D, Nordseth T, Loberg M, Skaug T, Bjornstad K, Gundersen O, Skjaervold NK, Klepstad P. Circulatory trajectories after out-of-hospital cardiac arrest: a prospective cohort study. BMC Anesthesiol. 2021 Sep 8;21(1):219. doi: 10.1186/s12871-021-01434-2. PMID 34496748
- [Result] Langeland H, Damas JK, Mollnes TE, Ludviksen JK, Ueland T, Michelsen AE, Loberg M, Bergum D, Nordseth T, Skjaervold NK, Klepstad P. The inflammatory response is related to circulatory failure after out-of-hospital cardiac arrest: A prospective cohort study. Resuscitation. 2022 Jan;170:115-125. doi: 10.1016/j.resuscitation.2021.11.026. Epub 2021 Nov 24. PMID 34838662
- [Derived] Farbu BH, Lydersen S, Mohus RM, Ueland T, Mollnes TE, Klepstad P, Langeland H. The detrimental effects of intestinal injury mediated by inflammation are limited in cardiac arrest patients: A prospective cohort study. Resusc Plus. 2024 Apr 17;18:100639. doi: 10.1016/j.resplu.2024.100639. eCollection 2024 Jun. PMID 38666252
- [Derived] Hoftun Farbu B, Langeland H, Ueland T, Michelsen AE, Jorstad Kruger A, Klepstad P, Nordseth T. Intestinal injury in cardiac arrest is associated with multiple organ dysfunction: A prospective cohort study. Resuscitation. 2023 Apr;185:109748. doi: 10.1016/j.resuscitation.2023.109748. Epub 2023 Feb 25. PMID 36842675
- [Derived] Langeland H, Bergum D, Loberg M, Bjornstad K, Skaug TR, Nordseth T, Klepstad P, Skjaervold NK. Characteristics of circulatory failure after out-of-hospital cardiac arrest: a prospective cohort study. Open Heart. 2022 Jan;9(1):e001890. doi: 10.1136/openhrt-2021-001890. PMID 35046124